CLINICAL TRIAL: NCT04096976
Title: Outcome After Near-Hanging Injury
Brief Title: Epidemiology and Determinants of Short-Term Outcome in Critically Ill Patients With Near-Hanging Injury
Acronym: ANTIGONE
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, LEGRIEL stephane, Principal Investigator, Versailles Hospital
Other Study IDs: P12/17_Antigone
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Near Hanging
MeSH Terms: interventions — Logistic Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital survival
  Interventions: Other: logistic regression
- No hospital survival
  Interventions: Other: logistic regression

INTERVENTIONS:
Other: logistic regression — To identify associations between factors listed in Table 1 and hospital survival, we used logistic regression

SUMMARY:
Near-Hanging is a catastrophic event that has been merely studied in the literature. We aimed to report the outcomes, and early predictors of hospital survivors in critically ill patients with near-hanging.

Patients admitted to 31 university or university-affiliated participating ICUs in France and Belgium between 1992 and 2014 were studied retrospectively. Hospital survival was the main judgment criterion.

ELIGIBILITY:
Inclusion Criteria:

* any of the following code corresponding in the International Statistical Classification of Diseases and Related Health Problems, 10th Revision: Intentional self-harm by hanging, strangulation and suffocation (X70). Local investigators reviewed the medical records of the patients thus identified to select adults admitted to the ICU after successfully resuscitated near-hanging injury.
* older than 18 years
* requiring ICU management

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult
Study Population: All eligible cases extracted from the participation ICUs hospital registries were included in the present study if they were older than 18 years, with in- or out-of-hospital near-hanging self-arm, and if they required ICU management.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 1992-01 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hospital survival | 1 year
  Survival rate at hospital discharge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Charentenay L, Schnell G, Pichon N, Schenck M, Cronier P, Perbet S, Lascarrou JB, Rossignol T, Lesieur O, Argaud L, Colin G, Cholley B, Quenot JP, Merdji H, Silva S, Piagnerelli M, Chelly J, Salvetti M, Couraud S, Deye N, Danguy des Deserts M, Paul M, Thiery G, Simon M, Martin C, Vincent F, Das V, Jacq G, Jacobs F, Soummer A, Mayaux J, Beuret P, Ouchenir A, Durant C, Darmon M, Azoulay E, Sauneuf B, Daubin C, Mongardon N, Biard L, Cariou A, Geeraerts T, Legriel S; Antigone Investigators. Outcomes in 886 Critically Ill Patients After Near-Hanging Injury. Chest. 2020 Dec;158(6):2404-2413. doi: 10.1016/j.chest.2020.07.064. Epub 2020 Aug 3. PMID 32758563